CLINICAL TRIAL: NCT00005100
Title: Measurement of Outcome of Surgical Treatment in Patients With Acromegaly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Columbia University (Other)
Other Study IDs: NCRR-M01RR00645-2525; CPMC-IRB-7590
Record Dates: First submitted 2000-04-06; First posted 2000-04-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Acromegaly
Keywords: acromegaly; endocrine disorders; rare disease
MeSH Terms: conditions — Acromegaly; Endocrine System Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Compare growth hormone (GH) levels at baseline and after glucose suppression measured with both a polyclonal radioimmunoassay and a highly sensitive immunoradiometric assay (IRMA) in patients with acromegaly and normal volunteers.

II. Measure the levels of IGF-I and its binding protein, IGFBP-3, in these cohorts.

III. Determine any correlation between levels of IGF-I and IGFBP-3 and GH suppressibility as assessed by sensitive IRMA.

IV. Determine if patients who demonstrate biochemical features of mild GH excess are at risk for progression to active disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Blood samples are collected and assessed for growth hormone and IGF-I by polyclonal radioimmunoassay (RIA) and immunoradiometric assay (IRMA). Growth hormone is measured at baseline and 60, 90, and 120 minutes after a 100 g glucose drink. Serum glucose is measured at baseline and at 2 hours post dextrose administration by the glucose hexokinase method.

Clinical scores are determined for headache, perspiration, fatigue, joint pain, and acne.

Exams and tests may be repeated every 6 months for 2 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of acromegaly and treated with transsphenoidal surgery

Biochemically and histologically confirmed growth hormone secreting tumor

OR

Healthy volunteers

--Prior/Concurrent Therapy--

Surgery:

* See Disease Characteristics
* Greater than 6 months since prior surgery

Other: At least 1 month since prior bromocriptine or octreotide

--Patient Characteristics--

Performance status: Ambulatory

Hepatic: No active hepatic disease

Renal: No active renal disease

Other:

* No diabetes mellitus
* No glucose intolerance
* Hypopituitarism allowed if on stable doses of replacement therapy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165
Dates: Start 1999-09

CONTACTS AND LOCATIONS:
Overall Officials: Pamela U. Freda, Study Chair — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States